CLINICAL TRIAL: NCT03073837
Title: RUDOLPH Study Nasal Microbiota and Concurrent Nose Soreness Associated With Common Cold Infection - a Pilot Using the HRV-16 Challenge Model in Healthy Subjects
Brief Title: Rudolph: Nasal Microbiota With Red and Sore Nose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kimberly-Clark Corporation (Industry)
Collaborators: NIZO Food Research (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 500-16-0006
Record Dates: First submitted 2017-02-21; First posted 2017-03-08 (Actual); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Dermatitis
MeSH Terms: conditions — Dermatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rhinovirus Challenge (Other): Challenge with HRV-16
  Interventions: Other: Rhinovirus Challenge

INTERVENTIONS:
Other: Rhinovirus Challenge — Challenge with HRV-16 virus

SUMMARY:
This pilot study will utilize the experimental rhinovirus infection model to study changes in skin microbiota in relation to skin erythema and soreness.

ELIGIBILITY:
Inclusion Criteria:

* self reported proneness to developing symptoms of nose redness and/or soreness
* sero-negative to HRV-16 at screening

Exclusion Criteria:

* confirmed or self-reported allergic rhinitis
* history of nasal or otologic surgery
* use of anti-inflammatory medication, recent antibiotics or anti-histamines

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2017-04-18 (Actual); Study Completion 2017-08-15 (Actual)

PRIMARY OUTCOMES:
nasal microbiota composition and occurrence of nose redness and soreness during rhinovirus infection | change from baseline compared to day 22
  Taxonomic classification of bacterial strains before and after HRV-16 virus for subjects with a VAS score rating >37mm

CONTACTS AND LOCATIONS:
Overall Officials: Lutter Rene, PhD, Principal Investigator — AIDS Malignancy Consortium
Locations (1):
- Academic Medical Center, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No